CLINICAL TRIAL: NCT02166957
Title: Evaluation of the Effectiveness of Endoscopic "Rendez-vous" Technique for Esophageal Reconstructions for the Treatment of a Total and Extensive Disruption of the Esophagus
Brief Title: Evaluation of the Effectiveness of Endoscopic "Rendez-vous" Technique Foresophageal Reconstructions for the Treatment of a Total and Extensive Disruption of the Esophagus
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, MD, Société Française d'Endoscopie Digestive
Other Study IDs: OESORDV; OESORECO
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Esophageal Disruption; Esophageal Obstruction
Keywords: Esophageal disruption; anterograde-retrograde endoscopy; rendez-vous technique; NOTES; recanalization; dilatations; Stenting; radiation therapy; head and neck carcinoma
MeSH Terms: conditions — Airway Obstruction; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Long disruption > 5cm +/- loss of SES
  Interventions: Procedure: Recanalization
- Short disruption < 5cm
  Interventions: Procedure: Recanalization

INTERVENTIONS:
Procedure: Recanalization — All patients received clear and detailed information about the different steps, the benefits and the risks of the procedure they would undergo, and gave an informed consent.
  The rendez-vous technique shared some common characteristics whatever the etiology and the length of esophageal disruption. First, prior to start the specific endoscopic management, all the patients needed to have undergone a surgical gastrostomy one month earlier in order to allow the retrograde access. This one-month delay was necessary to get it completely healed before using it for the procedure.
  The principle of the combined anterograde retrograde approach is to get an endoscopic access to both the proximal and distal side of the obstruction in the purpose to achieve better and safer recanalization, which could be carried out with either transillumination or using a needle under x-rays guidance.

SUMMARY:
Complete esophageal obstructions leads to definitive fasting. The rendez-vous endoscopic approach had already been described for complex stenoses but never for disruption with loss of tissue and SES. Patients and methods: This is a retrospective observationnal study about patients referred for complete esophageal disruption and classified in two groups: 1/ Long disruption (> 5cm), after caustic ingestion or due to an esophageal stripping during SEMS removal; 2/ Short disruption (< 5cm), consecutive to radiation therapy. All the procedures are performed according the anterograde retrograde approach, using CO2 and under X-rays guidance. We report the characteristeristics of the procedures, the efficacy, the time before discharge and refeeding, the complications, and the follow-up, especially the number of dilatation sessions for each group. The hypothesis is that anterograde retrograde endoscopic technique is safe and effective for the management of esophageal disruptions in patients for which the surgical treatment confers a high risk of morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal disruption with or without loss of SES

Exclusion Criteria:

* Esophageal Complex stenosis
* Mediastinitis
* Severe sepsis
* Coagulation abnormalities
* Contra-indications to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective report about six patients referred for complete esophageal disruption
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the rendez vous approach for treating esophageal disruption | 2 days
  We evaluate the technical and the clinical success. The technical success is the ability to recanalize the esophagus endoscopically.
  The clnical success is the possibility to feed patients.

SECONDARY OUTCOMES:
Number of endoscopic sessions | Up to 2 years
Time before refeeding | 15 days
Complications | 7 days
  Per-operative complications (bleeding, perforations, anesthesiological) and post-operative (infection, bleeding...)
Number of endoscopic dilation sessions after recanalization | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- APHM, North Hospital, Department of gastroenterology, Marseille, France